CLINICAL TRIAL: NCT01081925
Title: Congestive Heart Failure: Causes of Sudden Worsening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Pelouch Radek, MD, University Hospital Hradec Kralove
Other Study IDs: MSM0021620817-HKJC
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-02

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Cardiac Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Congestive heart failure: Patients suffering from sudden worsening of congestive heart failure

SUMMARY:
The purpose of the study is to recognize main causes of acute decompensation of chronic congestive heart failure.

DETAILED DESCRIPTION:
Congestive heart failure (CHF) presents a very significant cause of morbidity and mortality. The prevalence of CHF is between 2 and 4% and rises with age (in 70- to 80-year-old people is between 10 and 20%). CHF is the cause of 5% of all acute hospital admissions and accounts for 2% of expenses on health. The most common causes of worsening of the chronic CHF are ischemia, arrhythmias, valvular dysfunction, systemic or pulmonary hypertension, volume overload or fluid retention, high output conditions (infection, anemia, thyrotoxicosis), drugs (NSAIDs, cyclo-oxygenase (COX) inhibitors, thiazolidinediones) and medication nonadherence. The goal of this study is to determine the proportion of various reasons of acute worsening of CHF, using commonly available methods including assessment of serum drug levels.

ELIGIBILITY:
Inclusion Criteria:

* able to provide informed consent
* aged 19 years or more
* history of heart failure of at least one month
* examined or hospitalized for acute dyspnea at rest or with minimal exertion
* clinical signs of fluid overload defined as at least one of following:
* rales
* jugular venous distension
* peripheral edema
* pulmonary congestion on X-ray
* NT-proBNP above 210 pmo/l

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from sudden worsening of congestive heart failure, who are examined at the Emergency department or admitted to University Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Radek Pelouch, MD, Principal Investigator — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia